CLINICAL TRIAL: NCT01951781
Title: Rapid Quantitative Neutrophil CD64 Measurement for Early Diagnosis of Nosocomial Infection in Preterm Newborns
Brief Title: Neutrophil CD64 for Early Diagnosis of Nosocomial Infection in Preterm Newborns
Acronym: NEOCD64
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 9117
Record Dates: First submitted 2013-09-18; First posted 2013-09-27 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2013-09

CONDITIONS: Nosocomial Infection
Keywords: marker CD64; blood sample; nosocomial infection; preterm newborn
MeSH Terms: conditions — Cross Infection | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NEOCD64 (Other): NEOCD64 : dosage of CD64 blood marker in preterm newborn who are suspected of nosocomial infection (blood sample)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — blood sample in newborn preterms suspected of nosocomial infection (neoCD64 arm)
  When late-onset sepsis is suspected, blood samples are obtained from peripheral veins for a complete blood count, measurement of CRP and PCT concentration and one bacterial culture acording to the current recommendation of the CDC. CD64 concentration measurement require 0.2 ml aditionnal blood.

SUMMARY:
Diagnosis of late-onset sepsis is difficult in the absence of specific clinical signs and biological markers in the infection initial phase .The aim of this study is to determine the performance of a new infection marker : Neutrophil CD64 for early diagnosis in nosocomial infection (NI) in preterm newborns.

METHODS :

* Monocentric prospective study including preterm newborn infants (<37 weeks of gestationnal age ) with clinical suspicion of nosocomial infection in a neonatal intensice care unit (Neonatal intensive care unit of Montpellier, France).
* Patients will be enrolled in the study after informed consents. Rapid and automated CD64 measurment will be realized during the conventional blood sample including C-Reactive Protein (CRP), Procalcitonin (PCT) and blood culture.
* Broad-spectrum antibiotic therapy can be started on the advice of clinician and blinded the result of CD64. Patients will be then classed in three groups using CDC criteria (center for disease control) : 1-no infection, 2-infection, 3-possible infection during the multidisciplinary staff. Specificity, sensitivity, negative and positive value of CD64 will be calculated and the performances of CRP, PCT and CD64 will be compared.

  153 patients are needed in the study enrolled during a period of 12 months.

PERSPECTIVES Neutrophil CD64 monitoring might be help clinicians to manage nosocomial infections in neonates.CD64 allow to integrate in a decision algorithm with the determination of the best cut-off value to faster processing nosocomial infections and could help to reduce unnecessary antibioc therapy. A rapid technique for determination of CD64 should be readily available in our unit.

ELIGIBILITY:
Inclusion Criteria:

* preterm newborn (<37 weeks of gestationnal age )
* undergoing symptoms of late-onset-sepsis
* written informed consent obtained from the parents

Exclusion Criteria:

* patient undergoing antibiotic therapy
* patient undergoing surgery in the last seven days,
* patient with severe congenital malformation
* necrotizing enterocolitis
* parents unable to understand the purpose of the study
* no affiliation to social security

Max Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
proportion of negatives (healthy patient) which are correctly identified as such | day 1

SECONDARY OUTCOMES:
proportion of positives (sikness)which are correctly defined as such | day 1
  sensibility of CD64 value
negative predictive CD64 value | day 1
positive predictiveCD64 value | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Gilles CAMBONIE, Professor, Principal Investigator — Montpellier hospital
Locations (1):
- Montpellier University hospital, Montpellier, France